CLINICAL TRIAL: NCT06985602
Title: Adebrelimab Combined With Chemoradiotherapy Followed by Surgery for Locally Advanced or Limited Metastatic Gastric/ Esophagogastric Junction Adenocarcinoma.
Brief Title: Adebrelimab With Chemoradiotherapy and Surgery for G/GEJ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Cheng Chen, Doctor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAS-Jiangsu03
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal Adenocarcinoma; Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Adebrelimab Combined with Chemoradiotherapy Followed by Surgery (Experimental)
  Interventions: Combination Product: Arm 1: Adebrelimab Combined with Chemoradiotherapy Followed by Surgery

INTERVENTIONS:
Combination Product: Arm 1: Adebrelimab Combined with Chemoradiotherapy Followed by Surgery — * Adebrelimab: Given concurrently with chemotherapy, 1200mg by intravenous infusion every three weeks for four cycles.
  * Chemotherapy: Oxaliplatin 130mg/m² on day 1 + Capecitabine 1000mg/m² bid (XELOX regimen), from day 1 to day 14, repeated every three weeks for four cycles;
  * Radiotherapy: Unresectable limited metastatic lesions with SBRT; Potentially resectable lesions with low-dose radiotherapy.
  * Surgery: Performed 3-5 weeks after the completion of conversion therapy.

SUMMARY:
Gastric cancer is one of the most common and deadly cancers globally, characterized by a poor prognosis. Approximately 70% of patients are diagnosed at an advanced stage, and the 5-year survival rate is only around 10%. While advancements in targeted therapies and immunotherapy have improved treatment efficacy and extended survival, advanced gastric and gastroesophageal junction adenocarcinomas remain incurable. Subgroup analyses indicate that patients with limited metastases, such as liver oligometastasis or retroperitoneal lymph node metastasis, may benefit more from conversion therapy. However, current guidelines do not recommend specific treatment protocols for gastric cancer with limited metastasis. Immunotherapy has shown moderate efficacy in selected patients with advanced gastric adenocarcinoma. Additionally, low-dose radiotherapy (LDRT) may synergistically enhance antitumor responses when combined with immunotherapy. This Phase II trial aims to evaluate the safety and efficacy of combining Adebrelimab, chemotherapy, and LDRT before surgery in treating adult patients with gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed esophagogastric junction (EGJ)/gastric adenocarcinoma.
2. Patients with locally advanced disease (AJCC staging T4b or N2 fusion metastasis) or limited metastasis confirmed by endoscopy, CT, MRI, or PET/CT scans, and multidisciplinary team (MDT) discussion.
3. From a medical and surgical technical perspective, the primary lesion and surrounding abdominal lymph nodes are assessed as potentially resectable; limited metastatic lesions are evaluated by MDT for resectability or for the possibility of achieving curative treatment through other local treatment methods (such as local radiotherapy or radiofrequency ablation).
4. Exclusion of peritoneal metastasis.
5. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
6. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
7. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
8. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
9. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
10. Male or female. Age ≥ 18 years and ≤80 years.
11. Written (signed) informed consent.
12. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
13. Female patients should not be pregnant or breast feeding.

Exclusion Criteria:

1. Non-adenocarcinoma histology of gastric/esophagogastric junction tumors, such as squamous cell carcinoma or neuroendocrine carcinoma.
2. The primary lesion is considered unresectable from a medical or surgical technical perspective.
3. Imaging diagnosis indicates widespread metastasis (metastasis that does not meet the criteria for limited metastasis as defined above is considered widespread metastasis).
4. Peripheral neuropathy of grade ≥2.
5. Poor nutritional status, BMI <18.5 kg/m², or PG-SGA score ≥9.
6. Underwent major surgery or suffered a severe injury within 4 weeks prior to the first dose of the investigational drug.
7. Presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Received any investigational drug within 4 weeks prior to the first dose of the study drug.
9. Required systemic treatment with corticosteroids (daily >10 mg prednisone equivalent) or other immunosuppressive agents within 2 weeks prior to the first dose of the investigational drug.
10. Received an anti-tumor vaccine or live vaccine within 4 weeks before the first dose of the study drug.
11. Diagnosed with any active autoimmune disease or a history of autoimmune diseases.
12. History of immunodeficiency, including a positive HIV test, any acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation.
13. Any condition within 14 days prior to treatment requiring systemic corticosteroid therapy (dose>10mg/day of prednisone or equivalent) or other immunosuppressive treatments.
14. Presence of uncontrolled cardiac symptoms or conditions, such as:

    * NYHA Class II or higher heart failure
    * Unstable angina
    * Myocardial infarction within the past year
    * Clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
15. Severe infection within 4 weeks prior to the first dose, including pneumonia requiring hospitalization, bacteremia, or infectious complications.
16. History of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute pulmonary diseases.
17. Active pulmonary tuberculosis infection diagnosed by history or CT scan, or a history of active tuberculosis infection within the past year, or a history of untreated active tuberculosis infection more than one year ago.
18. Active hepatitis B or hepatitis C.
19. Laboratory abnormalities of sodium, potassium, or calcium greater than Grade 1 within 2 weeks before enrollment that cannot be corrected with treatment.
20. Known allergy to monoclonal antibodies, any PD-1 components, paclitaxel, capecitabine, or any components used in their formulations.
21. Pregnant or breastfeeding women, or women of childbearing potential who are unwilling or unable to use effective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Safety | From enrollment until the end of treatment, assessed up to 18 months.
  Treatment-related adverse events will be categorized by severity and relationship to treatment. Descriptive statistics will be used to summarize the frequency and types.

SECONDARY OUTCOMES:
R0 Rate | From the completion of conversion therapy until surgery, assessed within 8 weeks.. following treatment completion
  Defined as the proportion of patients who achieve complete resection with no tumor within 1 mm of the resection margins (R0), calculated by dividing the number of patients achieving R0 resection by the total number of evaluable patients.
Pathologic complete response | From the completion of conversion therapy until surgery, assessed within 8 weeks following treatment completion
  Defined as pT0N0M0
Progression-Free Survival | From enrollment until tumor progression or death from any cause, whichever occurs first, assessed up to 2 years
  Progression will be assessed based on imaging studies and clinical evaluation, using RECIST v1.1 criteria. Data will be summarized using Kaplan-Meier estimates, and hazard ratios will be calculated.
Overall Survival | From enrollment until death from any cause, assessed up to 3 years.
  Overall Survival will be assessed using Kaplan-Meier estimates. Median survival and survival rates at specific time points will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Chen, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu cancer hospital, Nanjing, Province, China

IPD SHARING:
Plan to Share IPD: Undecided